CLINICAL TRIAL: NCT05939700
Title: Mavacamten Pregnancy Surveillance Program
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV027-014
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Breastfeeding; Hypertrophic Cardiomyopathy; Pregnancy Related
MeSH Terms: conditions — Breast Feeding; Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Cohort 1: Pregnant or breastfeeding women exposed to mavacamten
  Interventions: Drug: Mavacamten

INTERVENTIONS:
Drug: Mavacamten — Observational study of individuals exposed to at least 1 dose of mavacamten at any time during pregnancy and/or breastfeeding

SUMMARY:
The purpose of this observational pregnancy safety study is to assess maternal, fetal, and infant outcomes after exposure to mavacamten at any time during pregnancy and/or breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Exposure to at least 1 dose of mavacamten at any time during pregnancy (from 4 months prior to conception to pregnancy outcome) and/or at any time during breastfeeding (up to 12 months of infant age or weaning, whichever comes first)
* At least 15 years of age or older at the time of enrollment
* Informed consent or institutional review board/ethics committee-approved waiver of informed consent

Exclusion Criteria:

- None

Min Age: 15 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Individuals 15 years of age or older who are exposed to at least 1 dose of mavacamten at any time during pregnancy and/or breastfeeding.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Pregnancy outcomes | Up to 10 months
  (1) Number of live births, full term or preterm births, stillbirths, spontaneous abortions, and elective abortions, (2) Number of participants with pregnancy complications
Fetal/neonatal/infant outcomes | Up to 12 months post pregnancy outcome
  Number of fetal/neonatal/infants in utero, at birth, and through the first year of life with major and minor congenital malformations, small for gestational age, premature delivery, and post-natal growth and development deficiency

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- The Mavacamten Pregnancy Surveillance Program, PPD Inc, Wilmington, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm